CLINICAL TRIAL: NCT00066066
Title: Effect of Three Periodontal Therapies in Current Smokers and Non-Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Forsyth Institute (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDCR-14242; R01DE014242 (NIH)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-03

CONDITIONS: Periodontitis; Periodontal Diseases
MeSH Terms: conditions — Periodontitis; Periodontal Diseases | interventions — Tooth Exfoliation; Root Planing; Metronidazole; Amoxicillin; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Scaling and root planing alone (Placebo Comparator): Full mouth scaling and root planing (SRP) alone plus a placebo pill taken twice daily for 2 weeks.
  Interventions: Procedure: Scaling and root planing
- SRP + Metronidazole (Active Comparator): Full mouth Scaling and Root Planing plus Metronidazole (MET) 250 mg tid x 14 days
  Interventions: Drug: Metronidazole
- SRP + MET + Amoxicillin + Doxycycline (Active Comparator): Full mouth Scaling and Root Planing plus Metronidazole (MET) 250 mg tid x 14 d and Amoxicillin (AMOX) 500 mg tid for 14 days and local drug delivery of Doxycycline (TET LDD) in pockets >4mm
  Interventions: Drug: Amoxicillin; Drug: Doxycycline

INTERVENTIONS:
Procedure: Scaling and root planing — Scaling and root planning (SRP) is the mechanical debridement of the tooth and root surfaces and is standard of care in periodontal therapy.
  Arms: Scaling and root planing alone
Drug: Metronidazole — Metronidazole (MET) is an antibiotic that is particularly effective against Gram negative bacterial species. The dose for this study is: 250 mg tid x 14d.
  Arms: SRP + Metronidazole
Drug: Amoxicillin — Amoxicillin (AMOX) is a broad spectrum antibiotic and was prescribed at 500 mg tid for 14d.
  Arms: SRP + MET + Amoxicillin + Doxycycline
Drug: Doxycycline — The ATRIDOX (doxycycline hyclate) ® product is a subgingival controlled-release product composed of a two syringe mixing system. Syringe A contains 450 mg of the ATRIGEL® Delivery System, which is a bioabsorbable, flowable polymeric formulation composed of 36.7% poly(DLlactide) (PLA) dissolved in 63.3% N-methyl-2-pyrrolidone (NMP). Syringe B contains 50 mg of doxycycline hyclate which is equivalent to 42.5 mg doxycycline. The constituted product is a pale yellow to yellow viscous liquid with a concentration of 10% of doxycycline hyclate. Upon contact with the crevicular fluid, the liquid product solidifies and then allows for controlled release of drug for a period of 7 days. Doxycycline is a broad-spectrum antibiotic synthetically derived from oxytetracycline.
  Other Names: Atridox
  Arms: SRP + MET + Amoxicillin + Doxycycline

SUMMARY:
The purpose of this study is to determine in current and non-smokers the clinical and microbiological effects of 3 therapies: scaling and root planing (SRP) alone; SRP in combination with the orally administered antibiotic metronidazole; and SRP with the orally administered antibiotics metronidazole and amoxicillin along with the locally delivered antibiotic doxycycline at periodontal pockets >= 4 mm.

DETAILED DESCRIPTION:
Cigarette smokers have more severe periodontal disease and more widespread colonization by periodontal pathogens than non smokers. In addition, smokers respond less well to periodontal therapies, particularly mechanical therapies such as scaling and root planing (SRP) and surgery. Recent data from our laboratory have indicated that treatment that included antibiotics produced a better clinical effect in smokers than mechanical therapy alone. Thus, the purpose of the present investigation is to compare the immediate and long-term effects of 3 periodontal therapies on clinical, microbiological and host parameters in current and non smokers. In this double blind, placebo-controlled, randomized study, 108 current smokers and 108 non smokers will be randomly assigned to 1 of 3 treatment groups: SRP alone; SRP + systemically administered metronidazole; SRP + systemically administered amoxicillin and metronidazole and local delivery of doxycycline at pockets > 4 mm. Plaque Index, Gingival Index, % of sites with bleeding on probing, suppuration, pocket depth and attachment level will be measured at 6 sites per tooth at all teeth excluding 3rd molars at baseline, 3, 6, 12, 18 and 24 months. Subgingival plaque samples taken from the mesial aspect of each tooth at the same time points will be analyzed individually for their content of 40 subgingival species using checkerboard DNA-DNA hybridization. Antibody levels to 20 subgingival species will be measured in serum samples taken at baseline, 6 and 24 months. Levels of IL-1b, IL-10 and IFNg will be measured in GCF samples taken from the 4 deepest pockets at baseline, 3, 6 and 24 months. The major hypothesis to be tested is whether smokers respond better to periodontal therapies that include 1 or more antibiotics. Other hypotheses will test whether host and microbiological parameters differ between smokers and non smokers and if such parameters are comparably altered after therapy in both groups. The results will be of immediate clinical benefit to the large segment of periodontal patients who smoke cigarettes. Smokers make up 26 - 30% of the adult population and form a disproportionately high segment of the population requiring periodontal treatment. They may have special needs in terms of periodontal therapy which should be clarified by the proposed investigation. In addition, the cigarette smoker is an example of a periodontal patient who is "compromised" in terms of his/her ability to cope with infectious diseases. The proposed investigation should provide a model to examine methods that could be useful in treating compromised patients whether compromised by harmful habits such as smoking, systemic disease or genetic background.

ELIGIBILITY:
Inclusion Criteria:

* > 20 teeth
* > 5% sites (approx. 8 sites) with pocket depth > 4 mm and / or 5% sites with attachment level > 4 mm and mean AL < 4.5 mm and mean PD < 3.9 mm (not including tooth brush abrasions).

Exclusion Criteria:

* > 50% of sites with pocket depth or attachment level > 4 mm
* Pregnancy or nursing
* Periodontal or antibiotic therapy in the previous 6 months
* Any systemic condition which might influence the course of periodontal disease or treatment (e.g. diabetes, AIDS)
* Any systemic condition which requires antibiotic coverage for routine periodontal procedures (e.g. heart conditions, joint replacements etc.)
* Liver disease
* Any known allergy to amoxicillin, metronidazole or doxycycline
* Lactose intolerance

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2003-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Haffajee, DDS, Principal Investigator — Boston, MA; Ricardo Teles, DDS, DMSc, Principal Investigator — The Forsyth Institute
Locations (1):
- Department of Periodontology, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Khattri S, Kumbargere Nagraj S, Arora A, Eachempati P, Kusum CK, Bhat KG, Johnson TM, Lodi G. Adjunctive systemic antimicrobials for the non-surgical treatment of periodontitis. Cochrane Database Syst Rev. 2020 Nov 16;11(11):CD012568. doi: 10.1002/14651858.CD012568.pub2. PMID 33197289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with moderate to advanced chronic periodontitis were recruited to the clinical center at The Forsyth Institute. Subjects were recruited from the Boston area, subjects of any racial / ethnic group were accepted for study.
Pre-assignment Details: Only 5 subjects dropped prior to randomization due to conflicts in scheduling or unable to adhere to the monitoring plan.
Groups:
- Scaling and Root Planing (SRP) Only NonSmokers; SRP Only Smokers: Subjects received full mouth scaling and root planing (SRP) under local anesthesia.Maintenance SRP was performed every 3 months for the duration of the study in all subjects.
- SRP and Metronidazole (MET) NonSmokers; SRP and Metronidazole (MET) Smokers: In addition to full mouth scaling and root planing under local anesthesia,subjects received systemically administered metronidazole (250 mg tid x 14 days). Maintenance SRP was performed every 3 months for the duration of the study in all subjects.
  Metronidazole is an antibiotic that is particularly effective against Gram negative bacterial species.
- SRP and Amoxicillin, MET, Local Tetracycline NonSmokers; SRP and Amoxicillin, MET, Local Tetracycline Smokers: In addition to full mouth scaling and root planing under local anesthesia,subjects received systemically administered metronidazole (250 mg tid x 14 days) together with systemically administered amoxicillin (500 mg tid for 14 days) and local delivery of doxycycline (Atridox) at teeth with pockets > 4 mm. Maintenance SRP was performed every 3 months for the duration of the study in all subjects.
  Tetracycline : Tetracycline is an antibiotic that has proved effective in killing bacteria in the periodontal pocket when applied locally.
Period: Overall Study
Arm/Group | Scaling and Root Planing (SRP) Only NonSmokers | SRP Only Smokers | SRP and Metronidazole (MET) NonSmokers | SRP and Metronidazole (MET) Smokers | SRP and Amoxicillin, MET, Local Tetracycline NonSmokers | SRP and Amoxicillin, MET, Local Tetracycline Smokers
Started | 27 | 22 | 30 | 20 | 27 | 20
Baseline | 27 | 22 | 30 | 20 | 27 | 20
3 Month | 21 | 17 | 23 | 16 | 22 | 15
6 Month | 19 | 13 | 23 | 13 | 21 | 14
12 Month | 18 | 11 | 21 | 11 | 19 | 9
Completed | 21 (27 enrolled, 21 analyzed,18 subjects had complete data,3 subjects had data carried forward.) | 18 (22 enrolled, 18 analyzed,11 subjects had complete data,7 subjects had data carried forward.) | 23 (30 enrolled, 23 analyzed,21 subjects had complete data,2 subjects had data carried forward.) | 16 (20 enrolled, 16 analyzed,11 subjects had complete data,5 subjects had data carried forward.) | 24 (27 enrolled, 24 analyzed,19 subjects had complete data,5 subjects had data carried forward.) | 15 (20 enrolled, 15 analyzed,9 subjects had complete data,6 subjects had data carried forward.)
Not Completed | 6 | 4 | 7 | 4 | 3 | 5
Not completed — Lost to Follow-up | 6 | 4 | 7 | 4 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Scaling and Root Planing (SRP) Only: Subjects received full mouth scaling and root planing (SRP) under local anesthesia.Maintenance SRP was performed every 3 months for the duration of the study in all subjects.
- SRP and Metronidazole (MET): In addition to full mouth scaling and root planing under local anesthesia,subjects received systemically administered metronidazole (250 mg tid x 14 days). Maintenance SRP was performed every 3 months for the duration of the study in all subjects.
  Metronidazole is an antibiotic that is particularly effective against Gram negative bacterial species.
- SRP and Amoxicillin, MET and Locally Delivered Tetracycline: In addition to full mouth scaling and root planing under local anesthesia,subjects received systemically administered metronidazole (250 mg tid x 14 days) together with systemically administered amoxicillin (500 mg tid for 14 days) and local delivery of doxycycline (Atridox) at teeth with pockets > 4 mm. Maintenance SRP was performed every 3 months for the duration of the study in all subjects.
  Tetracycline : Tetracycline is an antibiotic that has proved effective in killing bacteria in the periodontal pocket when applied locally.
- Total: Total of all reporting groups
Arm/Group | Scaling and Root Planing (SRP) Only | SRP and Metronidazole (MET) | SRP and Amoxicillin, MET and Locally Delivered Tetracycline | Total
Number analyzed (Participants) | 49 | 50 | 47 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 46 | 44 | 132
  >=65 years | 7 | 4 | 3 | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 50.3 (11.8) | 50.3 (11.6) | 48.0 (11.1) | 49.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 20 | 64
  Male | 28 | 27 | 27 | 82
Region of Enrollment [Number; unit: participants]
  United States | 49 | 50 | 47 | 146

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Clinical Attachment Level.
Description: Periodontal diseases are clinically diagnosed by assessments of gingival inflammation and measurements of tissue destruction. The damage to the apparatus of support of the teeth is quantified using measurements of probing pocket depth (PD) and clinical attachment level (CAL). These measurements are obtained using a periodontal probe which is introduced into the gingival sulcus to determine the distance in millimeters from the gingival margin to the depth of the sulcus or pocket (PD). Since the gingival margin fluctuates in response to inflammation (hyperplasia) or might recede, a more accurate measure of loss of attachment is obtained using the CAL, which measures the distance from a "fixed" landmark on the tooth such as the cemento-enamel junction to the depth of the pocket. Changes in CAL from baseline were used to assess results obtained with the treatment of periodontal diseases.
Time Frame: Baseline, 3, 6 and 12 months
Population: Of the 146 subjects, 117 were included in the analysis, who had 2 or fewer missing monitoring visits. 84 subjects had complete data, 23 subjects had one missing visit and 10 subjects had 2 missing visits. For the 33 subjects with missing visits, data were carried forward. 68 subjects were non smokers and 49 subjects were current smokers.
Measure: Mean (Standard Error); unit: mm
Groups:
- Scaling and Root Planing Only NonSmokers; SRP Only Smokers: Subjects received full mouth scaling and root planing (SRP) under local anesthesia.Maintenance SRP was performed every 3 months for the duration of the study in all subjects.
- SRP + Metronidazole NonSmokers; SRP + Metronidazole Smokers: In addition to full mouth scaling and root planing under local anesthesia,subjects received systemically administered metronidazole (250 mg tid x 14 days). Maintenance SRP was performed every 3 months for the duration of the study in all subjects.
  Metronidazole is an antibiotic that is particularly effective against Gram negative bacterial species.
- SRP + MET + Amoxicillin + Doxycycline NonSmokers; SRP + MET + Amoxicillin + Doxycycline Smokers: In addition to full mouth scaling and root planing under local anesthesia,subjects received systemically administered metronidazole (250 mg tid x 14 days) together with systemically administered amoxicillin (500 mg tid for 14 days) and local delivery of doxycycline (Atridox) at teeth with pockets > 4 mm. Maintenance SRP was performed every 3 months for the duration of the study in all subjects.
  Tetracycline : Tetracycline is an antibiotic that has proved effective in killing bacteria in the periodontal pocket when applied locally.
Arm/Group | Scaling and Root Planing Only NonSmokers | SRP Only Smokers | SRP + Metronidazole NonSmokers | SRP + Metronidazole Smokers | SRP + MET + Amoxicillin + Doxycycline NonSmokers | SRP + MET + Amoxicillin + Doxycycline Smokers
Number analyzed (Participants) | 21 | 18 | 23 | 16 | 24 | 15
mm
  Changes in mean CAL from baseline to 3 months | 0.11 (0.06) | 0.10 (0.04) | 0.21 (0.05) | 0.08 (0.06) | 0.29 (0.07) | 0.28 (0.06)
  Changes in mean CAL from baseline to 6 months | 0.15 (0.06) | 0.19 (0.05) | 0.19 (0.07) | 0.13 (0.07) | 0.34 (0.07) | 0.40 (0.08)
  Changes in mean CAL from baseline to 12 months | 0.11 (0.05) | 0.24 (0.05) | 0.26 (0.06) | 0.17 (0.09) | 0.41 (0.07) | 0.39 (0.08)
Statistical Analysis 1: Comparison: Scaling and Root Planing Only NonSmokers vs SRP + Metronidazole NonSmokers vs SRP + MET + Amoxicillin + Doxycycline NonSmokers; The null hypothesis of no difference among treatment groups in non-smokers was tested by comparing change in mean CAL in individuals at 3 months post-therapy; Test type: Superiority or Other; p > 0.05, ANOVA — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05
Statistical Analysis 2: Comparison: Scaling and Root Planing Only NonSmokers vs SRP + Metronidazole NonSmokers vs SRP + MET + Amoxicillin + Doxycycline NonSmokers; The null hypothesis of no difference among treatment groups in non-smokers was tested by comparing change in mean CAL in individuals at 6 months post-therapy; Test type: Superiority or Other; p > 0.05, ANOVA — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05
Statistical Analysis 3: Comparison: Scaling and Root Planing Only NonSmokers vs SRP + Metronidazole NonSmokers vs SRP + MET + Amoxicillin + Doxycycline NonSmokers; The null hypothesis of no difference among treatment groups in non-smokers was tested by comparing change in mean CAL in individuals at 12 months post-therapy; Test type: Superiority or Other; p < 0.05, ANOVA — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05
Statistical Analysis 4: Comparison: SRP Only Smokers vs SRP + Metronidazole Smokers vs SRP + MET + Amoxicillin + Doxycycline Smokers; The null hypothesis of no difference among treatment groups in smokers was tested by comparing change in mean CAL in individuals at 3 months post-therapy; Test type: Superiority or Other; p < 0.05, ANOVA — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05
Statistical Analysis 5: Comparison: SRP Only Smokers vs SRP + Metronidazole Smokers vs SRP + MET + Amoxicillin + Doxycycline Smokers; The null hypothesis of no difference among treatment groups in smokers was tested by comparing change in mean CAL in individuals at 6 months post-therapy; Test type: Superiority or Other; p < 0.05, ANOVA — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05
Statistical Analysis 6: Comparison: SRP Only Smokers vs SRP + Metronidazole Smokers vs SRP + MET + Amoxicillin + Doxycycline Smokers; The null hypothesis of no difference among treatment groups in smokers was tested by comparing change in mean CAL in individuals at 12 months post-therapy; Test type: Superiority or Other; p > 0.05, ANOVA — The p-value was not adjusted for multiple comparisons and the a priori threshold for significance was alpha = 0.05

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the entire course of the study for each enrolled subject.
Arm/Group | Scaling and Root Planing (SRP) Only NonSmokers | SRP Only Smokers | SRP and Metronidazole (MET) NonSmokers | SRP and Metronidazole (MET) Smokers | SRP and Amoxicillin, MET, Local Tetracycline NonSmokers | SRP and Amoxicillin, MET, Local Tetracycline Smokers
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/22 | 2/30 | 2/20 | 3/27 | 1/20
Other Adverse Events (participants affected / at risk) | 8/27 | 4/22 | 10/30 | 3/20 | 6/27 | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scaling and Root Planing (SRP) Only NonSmokers (N=27) | SRP Only Smokers (N=22) | SRP and Metronidazole (MET) NonSmokers (N=30) | SRP and Metronidazole (MET) Smokers (N=20) | SRP and Amoxicillin, MET, Local Tetracycline NonSmokers (N=27) | SRP and Amoxicillin, MET, Local Tetracycline Smokers (N=20)
hospitalizations (Surgical and medical procedures) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — One death was due to cancer - SRP/MET/NonSmoker Group One death due to unknown causes
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scaling and Root Planing (SRP) Only NonSmokers (N=27) | SRP Only Smokers (N=22) | SRP and Metronidazole (MET) NonSmokers (N=30) | SRP and Metronidazole (MET) Smokers (N=20) | SRP and Amoxicillin, MET, Local Tetracycline NonSmokers (N=27) | SRP and Amoxicillin, MET, Local Tetracycline Smokers (N=20)
Gastrointestinal Upset (Gastrointestinal disorders) | 8 (8) | 4 (4) | 10 (10) | 3 (3) | 6 (6) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes